CLINICAL TRIAL: NCT01234493
Title: Syndesmotic Injury and Fixation in SE Ankle Fractures: A Prospective Randomized Study
Brief Title: Syndesmotic Injury and Fixation in Supination-External (SE) Ankle Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Harri Pakarinen, Orthopedic surgeon, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SE4rand1
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Trauma
Keywords: ankle; fracture; syndesmosis;
MeSH Terms: conditions — Wounds and Injuries; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fixation (Active Comparator): Syndesmosis fixation with one 3.5mm fully threaded screw
  Interventions: Procedure: fixation
- no fixation (Active Comparator): No syndesmosis fixation
  Interventions: Procedure: no fixation

INTERVENTIONS:
Procedure: fixation — Syndesmosis fixation with one 3.5mm fully threaded three cortical screw
  Arms: fixation
Procedure: no fixation — No syndesmosis fixation.
  Arms: no fixation

SUMMARY:
The aim of our study was to determine whether transfixation of unstable syndesmosis is necessary in supination-external rotation type ankle fractures. Our hypothesis was that syndesmotic ligaments heal at the proper length after malleolar reduction and that syndesmotic transfixation is not needed in supination-external rotation fracture types.

DETAILED DESCRIPTION:
A prospective randomized study comparing syndesmotic transfixation to no fixation in AO/OTA Weber B-type ankle fractures was designed. To show a clinically significant difference (Olerud-Molander ankle score 20%, standard deviation (SD) 24 points, from our previous study) between the groups, the sample size was estimated (α=0.05, β=0.2, 20% drop out) to be 30 patients per group.

All skeletally mature patients (≥16 years old) with a unilateral Lauge-Hansen supination-external rotation type 4 ankle fractures treated within one week after injury at our hospital were considered eligible for the present study. Exclusion criteria were bilateral ankle fractures, pathologic fractures, concomitant tibial shaft fractures, previous significant injury or a fracture of either ankle, significant peripheral neuropathy, soft tissue infection in the region on either injured ankle, or inability to complete the study protocol.

After bony fixation, the 7.5-Nm standardized external rotation (ER) stress test for both ankles was performed under fluoroscopy. A positive stress examination was defined as a difference of more than 2 mm side-to-side in the tibiotalar or tibiofibular clear spaces on mortise radiographs. If the stress test was positive, the patient was randomized to either syndesmotic transfixation with 3.5-mm tricortical screws or no syndesmotic fixation.

Clinical outcome was assessed using the Olerud-Molander scoring system, RAND 36-Item Health Survey, and Visual Analogue Scale (VAS) to measure pain and function after a minimum 1-year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All skeletally mature patients (≥16 years old) with a unilateral Lauge-Hansen supination-external rotation type 4 ankle fractures treated within one week after injury at our hospital

Exclusion Criteria:

* Bilateral ankle fractures, pathologic fractures, concomitant tibial shaft fractures, previous significant injury or a fracture of either ankle, significant peripheral neuropathy, soft tissue infection in the region on either injured ankle, or inability to complete the study protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Olerud-Molander score | minimum one year

CONTACTS AND LOCATIONS:
Overall Officials: Harri J Pakarinen, MD, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No